CLINICAL TRIAL: NCT05515913
Title: Assessment of Nutrient Profile, Nutritional Status, Development and Severity of Children With Autistic Spectrum Disorder in Comparison With Typically Developing Children in Addis Ababa, Ethiopia
Brief Title: Nutritional Status and ASD Severity of Autistic Spectrum Disorder Children in Addis Ababa, Ethiopia; Case Control Study
Acronym: ASD
Status: Completed | Type: Observational
Sponsor: Addis Ababa University (Other)
Responsible Party: Principal Investigator, Feven yirgu Tamire, Principal Investigator, Addis Ababa University
Other Study IDs: AASTUASD
Record Dates: First submitted 2022-08-19; First posted 2022-08-25 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Autistic Spectrum Disorder
Keywords: Autistic spectrum disorder (ASD); Typically developing children (TDC); Nutritional status; Nutrient intake; Urine Iodine; Autistic severity
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Nutritional Status; Eating; Nutrition Assessment

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ASD ( autistic spectrum disorder): Children already diagnosed with autistic spectrum disorder
  Interventions: Other: Nutritional status; Behavioral: Eating behavior; Other: Urine iodine concentration; Other: Nutrient intake; Other: Dietary assessment; Other: Childhood autism rating scale
- TDC (typically developing children): Children within the typically development
  Interventions: Other: Nutritional status; Other: Urine iodine concentration; Other: Nutrient intake; Other: Dietary assessment

INTERVENTIONS:
Other: Nutritional status — Nutritional status of children as analyzed by anthropometric indices was under study
Behavioral: Eating behavior — The eating behavior of ASD children as analyzed by frequency of refusal of new food, sensitivity to food, food allergy and gastrointestinal systems was under study
  Groups: ASD ( autistic spectrum disorder)
Other: Urine iodine concentration — the 24 urine iodine concentration of all subjects was under study
Other: Nutrient intake — The nutrient intake as analyzed by three days food diary and major meal proximate analysis of subjects was under study
Other: Dietary assessment — The food frequency and dietary diversity of all subjects as analyzed by food frequency questioner, dietary diversity score and food variety score was under study
Other: Childhood autism rating scale — The autistic severity of ASD diagnosed children was under study as analyzed by childhood autism rating scale diagnosis
  Groups: ASD ( autistic spectrum disorder)

SUMMARY:
The study conducts a case control analysis of the nutritional status and intake of autistic spectrum disorder diagnosed children as compared to typically developing children in Addis Ababa, Ethiopia. It included analysis of anthropometric measurements, three days food diary food intake, urinary iodine analysis, childhood autism rating scale diagnosis, food frequency and eating behavior questioner and proximate analysis of one day major meals of selected subjects.

DETAILED DESCRIPTION:
Sample population was Addis Ababa city in which subjects were selected from one of the two autism centers in the country. Random sampling method was applied to select subject from the total enrolled children in the center using Ryan 2013 sample size calculation formula.

Subjects already diagnose with autistic spectrum disorder that didn't have any other chronic disease that affect diet and nutrition were included in the study. Subjects were selected randomly from each grade level in the center. They were registered and taken for data collection. Sample and Data was collected with the help of each child's center caregiver and parent. Childhood autism rating scale diagnosis, eating behavior analysis were analyzed for the ASD and anthropometric indices Z scores, urine iodine concentration, three days food diary analysis, major meals proximate analysis, food frequency and dietary diversity was assessed and compared to typically developing children in Addis Ababa.

Data entry and analysis was conducted using Emergency Nutrition Assessment software, Microsoft excel and Statistical Package for the Social Sciences software.

ELIGIBILITY:
Inclusion Criteria:

* Children already diagnosed with ASD
* school aged children (4-18 years old)

Exclusion Criteria:

* children with chronic illnesses ( such as cancer..)
* children taking heavy medications that may affect diet and nutrition

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The target population of this study were school-aged (i.e. 4-17 years old) children with ASD residing in Addis Ababa, Ethiopia. The study was conducted in one of the two selected autism center in Addis Ababa Ethiopia , one of the two autism centers in Ethiopia. Controls were selected from typically developing children's population of the same area as of ASD population.
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2021-08-14 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2022-02-08 (Actual)

PRIMARY OUTCOMES:
Body Mass Index for age z-scores | 1 day
  Body Mass Index and age will be combined to report Body mass index for age z-score in Kg/m2 for age in months
Height for age z-scores | 1 day
  Height and age will be combined to report height for age z-scores in centimeter for age in months
Weight for age z-scores | 1 day
  weight and age will be combined to report weight for age z-scores in kg for age in months
Zinc intake using three days food diary questioner | 5 days
  Three days food diary questioner will be used to report intake of zinc in mg/day
Energy intake using three days food diary questioner | 5 days
  Three days food diary questioner will be used to report intake of energy in kcal/day
Protein intake using three days food diary questioner | 5 days
  Three days food diary questioner will be used to report intake of protein in gm/day
Lipid intake using three days food diary questioner | 5 days
  Three days food diary questioner will be used to report intake of lipid in gm/day
Carbohydrate intake using three days food diary questioner | 5 days
  Three days food diary questioner will be used to report intake of carbohydrate in gm/day
Calcium intake using three days food diary questioner | 5 days
  Three days food diary questioner will be used to report intake of calcium in mg/day
Iron intake using three days food diary questioner | 5 days
  Three days food diary questioner will be used to report intake of Iron in mg/day
Thiamine intake using three days food diary questioner | 5 days
  Three days food diary questioner will be used to report intake of Thiamine in mg/day
Vitamin C intake using three days food diary questioner | 5 days
  Three days food diary questioner will be used to report intake of vitamin C in mg/day
Vitamin B2 intake using three days food diary questioner | 5 days
  Three days food diary questioner will be used to report intake of vitamin B2 in mg/day
Niacin intake using three days food diary questioner | 5 days
  Three days food diary questioner will be used to report intake of niacin in mg/day
Vitamin A intake using three days food diary questioner | 5 days
  Three days food diary questioner will be used to report intake of vitamin A in mg/day
Urine iodine concentration of children | 2 month
  Urine iodine concentration of children in µg /L
Autism symptom severity of children using Childhood Autism rating Scale diagnosis | 2 days
  Childhood autism rating scale assessed by total raw scores by age. for age 0-12, scores of 15-29.5 indicate limited behavior related to autism, score of 30-36.5 indicate mild to moderate level of behavior related to autism, score 37-60 indicate sever level behavior related to autism. for age 13 years and older, 15-27.5 indicate limited behavior related to autism, score of 28-34.5 indicate mild to moderate level of behavior related to autism, score 35-60 indicate sever level behavior related to autism.

SECONDARY OUTCOMES:
energy intake using proximate analysis of one day major meals | 2 months
  proximate analysis of one day major meals will be used to report intake of energy in k cal /100gm
Ash intake using proximate analysis of one day major meals | 2 months
  proximate analysis of one day major meals will be used to report intake of Ash in gm/100gm
Lipid intake using proximate analysis of one day major meals | 2 months
  proximate analysis of one day major meals will be used to report intake of lipid in gm/100gm
protein intake using proximate analysis of one day major meals | 2 months
  proximate analysis of one day major meals will be used to report intake of protein in gm/100gm
Carbohydrate intake using proximate analysis of one day major meals | 1 week
  proximate analysis of one day major meals will be used to report intake of carbohydrate in gm/100gm
frequency of food group consumption using food frequency questioner | 5 days
  percentage of children consuming from each food groups using a food frequency questioner
dietary diversity score of children using three days food diary | 5 days
  consumption of 1-3 food groups is scored as low dietary diversity score, consumption of 4-5 food groups is scored as medium dietary diversity score, consumption of >5 food groups is scored as high dietary diversity score.
frequency of food refusal in children using a questioner | 5 days
  frequency is scored as never to seldom, mild and sever
frequency of sensitivity to food | 5 days
  frequency is scored as never to seldom, mild and sever
frequency of gastrointestinal symptoms | 5 days
  frequency is scored as never to seldom, mild and sever
frequency of food allergic reactions | 5 days
  frequency is scored as never to seldom, mild and sever

CONTACTS AND LOCATIONS:
Overall Officials: Feven Yirgu Tamire, Principal Investigator — Addis Ababa Science and Technology University
Locations (1):
- Addis Ababa Science and Technology University, Addis Ababa, Ethiopia

IPD SHARING:
Plan to Share IPD: Undecided
Due to Ethical issue, sharing data to 3rd party is not decided yet.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-19): https://cdn.clinicaltrials.gov/large-docs/13/NCT05515913/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-19): https://cdn.clinicaltrials.gov/large-docs/13/NCT05515913/ICF_001.pdf